CLINICAL TRIAL: NCT07280923
Title: Reliability and Validity of the Pressure Relief Frequency Scale
Brief Title: Reliability and Validity of the PReFS
Acronym: PReFS
Status: Recruiting | Type: Observational
Sponsor: Baylor University (Other)
Responsible Party: Sponsor
Other Study IDs: 2339946
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Neurologic Disorders; Spinal Cord Injury; Stroke; Traumatic Brain Injury
Keywords: wheelchair user; pressure relief; skin integrity
MeSH Terms: conditions — Nervous System Diseases; Spinal Cord Injuries; Stroke; Brain Injuries, Traumatic | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wheelchair Users: Individuals with a neurologic disorder who are primary wheelchair users
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Participants will be interviewed for this study. No intervention will occur.

SUMMARY:
This study is testing the psychometric properties of a new tool to determine recommendations for pressure relief frequency in wheelchair users.

DETAILED DESCRIPTION:
The goal of the proposed study is to establish the content validity and inter-rater reliability of a new tool, the Pressure Relief Frequency Scale (PReFS). Findings from this study will provide clinicians with a tool that can be used to develop an individualized approach to teaching patients how frequently to perform weight shifts. The part of the study will establish the inter-rater reliability of the PReFs through video recordings of individuals who are wheelchair users.

ELIGIBILITY:
Inclusion Criteria:

* primary wheelchair user
* diagnosed with a neurologic disorder

Exclusion Criteria:

* does not use a wheelchair for more than 50% of waking hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a diagnosed neurologic disorder who are primary wheelchair users.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Interview | Baseline
  Each participant will take part in a 10-minute interview to answer questions on the PReFS

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ardolino, PT, PhD, Principal Investigator — Baylor University
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided